CLINICAL TRIAL: NCT01883388
Title: Assessing the Ability of An Innovative Screening Method To Identify Proteomic Changes In Cancer Patients- Protocol
Brief Title: NovellusDx Cancer Early Detection Blood Test- Clinical Trial
Status: Completed | Type: Observational
Sponsor: Fore Biotherapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: RAM-NOVEL-211-2012
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2014-10

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; blood sample
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
NovellusDx early detection test is a simple to perform blood test, which identifies the deregulated signaling pathways within the patient tumor based on protein secretion to the blood, thus enabling early stage disease signature detection. The investigators' current clinical trial is focused on proving the main feature of NovellusDx's Early Detection Test- discriminating between cancer patients and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* subjects ages 18 and above ICF obtain

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and subjects with primary / relapsed lung cancer
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a significant cancer fingerprint as measured by NovellusDX Cancer Early Detection test | 3.5 years
  NovellusDX Cancer Early Detection test will identify participants with significant cancer fingerprint based on tumor protein secretion to the blood circulation in sick subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yishai Ofran, MD, Principal Investigator — Rambam MC. Haematology Department
Locations (1):
- Rambam MC, Haifa, Israel